CLINICAL TRIAL: NCT00859014
Title: Safety/Feasibility of Autologous Mononuclear Bone Marrow Cells in Stroke Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sean Savitz, Professor, Neurology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01-HB-37163-05; R21HD060978 (NIH)
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Bone Marrow Mononuclear Cells (Experimental): Harvest of bone marrow from ischemic stroke patients, isolation and purification of mono-nuclear cell fraction from bone marrow, intravenous administration of autologous bone marrow mono-nuclear cells with a targeted dose of 10 million cells / kg.
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Bone Marrow Mononuclear Cells — Harvest of bone marrow from ischemic stroke patients, isolation of bone marrow mono-nuclear cells, and peripheral IV infusion of autologous bone marrow mono-nuclear cells

SUMMARY:
The purpose of this research study is to find out if bone marrow treatment (bone marrow aspiration and infusion of stem cells) can be safely used in adults who have recently (within 24-72 hours)suffered an acute ischemic stroke.

DETAILED DESCRIPTION:
Our primary hypothesis is that autologous bone marrow mononuclear cell transplantation by intravenous administration is feasible and safe after acute ischemic stroke. Our secondary hypothesis is that autologous transplantation is associated with improved outcome after acute stroke.

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke
2. age 18 to 83 years If >80 then the pre-stroke mRS needs to be < 1)
3. Right hemisphere NIHSS 6 -15, left hemisphere NIHSS 6-18
4. known onset time of acute symptoms
5. stem cell transplantation procedure must be performed within 24 to 72 hrs after stroke symptom onset
6. TPA infusion is allowed

Exclusion Criteria:

1. NIHSS 1a > 1
2. pre-stroke mRS > 1 if > 80 years of age
3. Ischemic stroke in the last 3 months, any vascular territory
4. MI, primary hemorrhagic or traumatic lesion of the brain within the last 3 months or identified on MRI. Small hemorrhagic transformation of the acute infarct is allowed.
5. seizure disorder
6. developmental delay
7. chronic kidney disease defined as baseline creatinine >1.4
8. hepatic disease or altered liver function as defined by SGPT >150 U/L and or T. Bilirubin >1.6 mg/dL at admission
9. pulmonary disease (e.g, COPD with oxygen-requirement at rest or with ambulation, moderate to severe asthma)
10. mechanical heart valve
11. Active malignancy or diagnosis of malignancy within 5 years prior to the start of screening or any history of chemotherapy or radiation affecting the bone marrow. Skin cancers (except for melanoma) are permitted.
12. prior immunosuppression, including chemotherapy administration within last 3 years or current immunosuppression as defined by WBC <3 x 103 cells/ml
13. known HIV
14. hemoglobin <10g/dl
15. uncorrected coagulopathy at the time of consent defined as INR >1.4; PTT>37 sec, or thrombocytopenia (PLT<100,000)
16. any hemodynamic instability at the time of consent (e.g, requiring continuous fluid resuscitation or ionotropic support).
17. Hypoxemia (SaO2<90%) at the time of consent, respiratory distress or persistent hypoxemia defined as SaO2 <94% for >30 minutes occurring at any time from hospital admission to time of consent. Intubation alone is not an exclusion.
18. pregnancy or positive b-HCG
19. current participation in any interventional research study
20. unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation
21. Multiple anti-platelet medications (Aggrenox is considered a single platelet agent)
22. Unable to undergo MRI or CT scan
23. Any other condition that the investigator feels would pose a significant hazard to the patient if enrolled.
24. Exclude infarct lesion size >145cc unless the NIHSS 1a remains < 1 and there is no evidence of infarct expansion or edema formation on any imaging obtained from admission up to the point just prior to infusion.
25. Exclude IA therapy use or if there is a planned or anticipated hemicraniectomy. Diagnostic angiograms are allowed
26. CT and/or Multimodal MRI exclusion criteria will be:

    * hemispheric strokes < 1.5 cm maximum diameter (on the MRI as seen on the diffusion-weighted imaging or CT)
    * midline shift >1mm or significant hemorrhagic transformation of the acute infarct

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean I Savitz, MD, Principal Investigator — University of Texas Heath Science Center- Houston
Locations (1):
- Memorial Hermann Hospital-Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Vahidy FS, Alderman S, Savitz SI. Challenges enrolling patients with acute ischemic stroke into cell therapy trials. Stem Cells Dev. 2013 Jan 1;22(1):27-30. doi: 10.1089/scd.2012.0404. Epub 2012 Oct 15. PMID 22970907
- [Result] Savitz SI, Misra V, Kasam M, Juneja H, Cox CS Jr, Alderman S, Aisiku I, Kar S, Gee A, Grotta JC. Intravenous autologous bone marrow mononuclear cells for ischemic stroke. Ann Neurol. 2011 Jul;70(1):59-69. doi: 10.1002/ana.22458. PMID 21786299

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Bone Marrow Mononuclear Cells
Started | 25
Completed | 20
Not Completed | 5
Not completed — Death | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Total number of study participants
Arm/Group | Autologous Bone Marrow Mononuclear Cells
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (13.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Study Related Serious Adverse Events (SR-SAE)
Description: Study Related Serious Adverse Events (SAE) as adjudicated by the DSMB - "Events"
Time Frame: 2 Years
Measure: Number; unit: Events
Arm/Group | Autologous Bone Marrow Mononuclear Cells
Number analyzed (Participants) | 25
Events | 0

2. Secondary Outcome: Functional Outcome
Description: Modified Rankin Scale (mRS) Score. The mRS is a six point (scored: 0 - 5) scale that measures post stroke disability. A seventh category (mRS = 6) is for patients who have died. A higher score indicates greater degree of disability. Patients scoring '5' are bed ridden, where as those scoring '0' are completely symptom free and independent.
Time Frame: 90-days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Autologous Bone Marrow Mononuclear Cells
Number analyzed (Participants) | 25
units on a scale | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Autologous Bone Marrow Mononuclear Cells
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous Bone Marrow Mononuclear Cells (N=25)
Ischemic Stroke (Nervous system disorders) | 2 — Not Study Related
Myocardial Infarction (Cardiac disorders) | 1 — Not Study Related
Stroke Expansion (Nervous system disorders) | 3 — Not Study Related
Syncope (Nervous system disorders) | 2 — Not Study Related
Hypotension (Vascular disorders) | 1 — Not Study Related
Renal Failure (Renal and urinary disorders) | 3 — Not Study Related
Sepsis (Infections and infestations) | 1 — Not Study Related
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 — Not Study Related
Seizure (Nervous system disorders) | 2 — Not Study Related
Carotid Hyperperfusion Syndrome (Nervous system disorders) | 1 — Not Study Related
Primary Non Small Cell Lung Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Not Study Related
Congestive Heart Failure (Cardiac disorders) | 1 — Not Study Related
Urinary Tract Infection (Renal and urinary disorders) | 1 — Not Study Related
Bradycardia (Cardiac disorders) | 1 — Not Study Related
Fracture Lumbar Vertebra (Musculoskeletal and connective tissue disorders) | 1 — Not Study Related
Numbness (General disorders) | 1 — Not Study Related
Hypertension (Vascular disorders) | 1 — Not Study Related
Pyelonephritis (Renal and urinary disorders) | 1 — Not Study Related
Hospital admission for observation (General disorders) | 1 — Not Study Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous Bone Marrow Mononuclear Cells (N=25)
Anemia (Blood and lymphatic system disorders) | 5 — Not Study Related
Leukocytopenia (Blood and lymphatic system disorders) | 3 — Not Study Related
Pain (Musculoskeletal and connective tissue disorders) | 9 — Non-specific Musculoskeletal Pain
Colitis (Gastrointestinal disorders) | 2 — Not Study Related
Nausea (General disorders) | 2 — Not Study Related
Vomitting (General disorders) | 2
Culture Bottle Skin Contamination, Suspected (General disorders) | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 — Not Study Related. All occurred greater than 4 months after enrollment
Urinary Tract Infection (Infections and infestations) | 10 — Nine patients were foley catheter associated. Remaining (one) experienced symptoms prior to infusion
Fall (General disorders) | 2 — Not Study Related
Prolonged Partial Thromboplastin Time (Blood and lymphatic system disorders) | 3 — Not Study Related
Increased Alanine Aminotransferase (Investigations) | 7 — All events are grade 1. All patients were on statins. Three patients had transient increase within 30 days and resolved. Three patients continued to fluctuate beyond 30 days. Two patients had normal ALT up till 30 days and later had elevation
Increased Aspartate Aminotransferase (Investigations) | 11 — All events are grade 1. All patients were on statins. Five patients had transient increase within 30 days and resolved. Two patients continued to fluctuate beyond 30 days. Four patients had normal AST up till 30 days and later had elevation
Increased INR (Investigations) | 5 — Not Study Related
Increased Lipase (Investigations) | 2 — Adjudicated as statin related
Hyperglycemia (Investigations) | 6 — Not Study Related
Hypernatremia (Investigations) | 3 — Not Study Related
Hypoalbuminemia (Investigations) | 4 — Not Study Related
Hypocalcemia (Investigations) | 7 — Not Study Related
Hypokalemia (Investigations) | 3 — Not Study Related
Hyponatremia (Investigations) | 4 — Not Study Related
Hypophosphatemia (Investigations) | 3 — Not Study Related
Headache (General disorders) | 2 — Not Study Related
Hemorrhagic Transformation of Ischemic Stroke (Nervous system disorders) | 7 — All events are grade 1 and were asymptomatic.
Ischemic Stroke (Nervous system disorders) | 2 — All events are grade 1, were asymptomatic, and were not study related.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 — Not Study Related
Decubitus Ulcer (General disorders) | 3 — Not Study Related
Peripheral Edema (General disorders) | 3 — Not Study Related
Hypotension (Vascular disorders) | 5 — Four events were not study related. Remaining (one) was relative hypotension.
Decreased Hemoglobin (Blood and lymphatic system disorders) | 14 — Six Not Study Related. All events grade 1 and 2

LIMITATIONS AND CAVEATS:
This is a Phase I safety and feasibility study, designed without a control group. Small sample size and inclusion of selected patients warrants caution in interpretation of findings. A randomized controlled study is needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes